CLINICAL TRIAL: NCT05722769
Title: RCT to Evaluate Bystander-informed CSTOP Now! to Prevent Child Sex Trafficking in Kentucky Middle Schools
Brief Title: CSTOP Now! Child Sex Trafficking Stops With You
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann Coker (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ann Coker, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 77232; U01CE003394 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-02-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Child Sex Trafficking
Keywords: Prevention

STUDY DESIGN:
Intervention Model Description: Randomization at Kentucky County level. Schools in counties randomized to the intervention receive the online intervention training. Schools in counties randomized to the attention control receive the attention control training.
Masking Description: County-level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CSTOP Now! Child Sex Trafficking Stops with You (Experimental): For this RCT, our research team has created CSTOP Now! online, interactive learning management system training. This CSTOP Now! online training will be offer to middle school staff in Kentucky counties randomized to this experimental intervention arm. This training seeks to provide middle school staff with information and resources to identify, intervene in, and prevent child sex trafficking (CST). This training will provide middle school staff with the knowledge, skills, and efficacy to intervene with children at risk of or experiencing CST. This training will also provide staff with skills to disrupt harmful attitudes or misinformation about CST.
  Interventions: Behavioral: CSTOP Now!
- Prevent Child Abuse Kentucky Online Training (Active Comparator): With input from Prevent Child Abuse Kentucky, our team developed training delivered via LMS and designed to identify child sex trafficking among middle school students. Only for middle school staff in counties randomized to the active comparator, we offer this online training using the same approach as that for staff in the intervention condition.
  Interventions: Behavioral: Prevent Child Abuse Kentucky Online Training

INTERVENTIONS:
Behavioral: CSTOP Now! — Child sex trafficking stops with you. Implement and evaluate the effectiveness of a multi-level bystander-informed program (CSTOP Now!) aimed at Kentucky public middle school staff. Participants will be trained to use the See It To Stop It Indicator Tool (SITSII) by using tiers of concern (clear concern, possible concern, and monitor of emerging concern). The SITSII tool directs the bystander actions to Decide, Directly Intervene, Disrupt, Delegate, and Document.
  Arms: CSTOP Now! Child Sex Trafficking Stops with You
Behavioral: Prevent Child Abuse Kentucky Online Training — The Kentucky State Police, in association with Prevent Child Abuse Kentucky, have developed videos we invite active comparator schools to review which also include how to identify and report child sex trafficking.
  Arms: Prevent Child Abuse Kentucky Online Training

SUMMARY:
Focus: Intervention & prevention of child commercial sexual exploitation or trafficking (CST) In Kentucky, familial SU/D increases risk of CST.

Primary goal: Implement and evaluate effectiveness of multi-level bystander-informed program (CSTOP Now!) aimed at Kentucky public middle schools for staff.

DETAILED DESCRIPTION:
Randomization will occur at the Kentucky county level among 50 counties with at least 2 middle schools for a middle school-based cluster RCT set in 50 of Kentucky's 120 counties. Middle schools in half (n=25) of the 50 Kentucky counties will be randomized to the intervention condition, while middle schools in the remaining 25 Kentucky counties will be randomly assigned to the attention control. We have selected counties that are similar in population size, demographics (% white, % <18 years of age, and % living in poverty, using 2019 Census estimates). Within each county, all middle schools (>200 across 50 counties) will be invited to participate in this RCT.

Participating staff will be emailed a link that will take them to a description of the study. Participation will involve receipt of online training, as randomized at the county level, and completing surveys immediately before receipt of the first training and at the end of each of school terms annually.

Aim 1. Evaluate the effectiveness of child sex trafficking (CST) prevention training implemented among middle school staff randomized, at the Kentucky county level, to change middle school staff:

1. Knowledge of child sexual exploitation and trafficking (hypothesize greater knowledge in Intervention versus Control),
2. Attitudes towards child sexual exploitation and trafficking (hypothesize lower stigma in Intervention versus Control),
3. Willingness and efficacy to intervene (hypothesize greater efficacy in Intervention versus Control),
4. Use of 'bystander' actions to thwart child sexual exploitation and trafficking risk (hypothesize increase actions in Intervention versus Control),
5. Use child sex trafficking screening, referral and reporting (hypothesize increase actions in Intervention versus Control),

Aim 2. Evaluate effectiveness of child sex trafficking mass media intervention (Intervention versus Control), randomized and measured at the Kentucky county-level, based on middle school staff survey data:

1. To increase child sexual exploitation and trafficking screening & reporting in short term (Years 1-2),
2. Begin to reduce child sexual exploitation and trafficking rates in longer term (Year 3-4) Analyses for both aims will be adjusted for school and county-level attributes

ELIGIBILITY:
Inclusion Criteria:

* Kentucky middle school staff in a public school
* Kentucky middle school staff in the intervention or attention control schools/counties.

Exclusion Criteria:

* Kentucky middle school staff not in intervention or attention control schools/counties.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5408 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge and Attitudes toward Child Sex Trafficking (CST) among middle school staff | Year 2-Year 4
  Knowledge of CST to include legal and behavioral definitions, risk factors, signs and symptoms, and awareness CST in staff's school or community Attitudes toward CST include stereotypes of those trafficked, their families and consumers, staff's empathy and attitudes toward helping those trafficked, self-efficacy to address CST with students or staff.
  Sex Trafficking Attitudes Scale, Human Trafficking Myths Scale, Adaptation of Self-Confidence and Screening Behaviors for Domestic Violence Scale

SECONDARY OUTCOMES:
Use of bystander actions and See It To Stop It Indicator (SITSII) screening tool | Year 2-Year 4
  Use of active bystander behaviors to prevent or stop child sex trafficking.
  Bystander behaviors to include the number of events reported by middle school staff to include directly intervene, delegate, disrupt, and document of behaviors to prevent child sex trafficking or report potential child sex trafficking.
  Based on Banyard, Plante, Moynihan (2005) Bystander Efficacy Scale and adapted for child sex trafficking.

CONTACTS AND LOCATIONS:
Overall Officials: Ann L. Coker, PhD, MPH, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No